CLINICAL TRIAL: NCT04821401
Title: Rejuvant™ Safety and Biomarker Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ponce De Leon Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PDLH-2019-01
Record Dates: First submitted 2021-03-22; First posted 2021-03-29 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Aging Well

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled trial in adult men ages 45-75 years and postmenopausal women up to age 75 years
Who Masked: Participant, Care Provider, Investigator
Masking Description: The medical assistant conducting clinical visits will receive two binders with sets of sequentially numbered, Kit Assignment Forms (n = 50) - one binder for men and one binder for women. For each new participant, the assistant will enter the participant identification # on the next Kit Assignment Form which contains the Kit # to be assigned to the new participant. The kits (contain either the dietary supplement or the placebo) were assigned either dietary supplement or placebo per the order of the randomization list generated by www.randomization.com
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Males study product (Experimental): 25 men will be randomized to Rejuvant
  Interventions: Dietary Supplement: Rejuvant
- Males placebo (Placebo Comparator): 25 man will be randomized to placebo
  Interventions: Dietary Supplement: Placebo
- Females study product (Experimental): 25 women will be randomized to Rejuvant
  Interventions: Dietary Supplement: Rejuvant
- Females placebo (Placebo Comparator): 25 women will be randomized to placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Rejuvant — Rejuvant tablets are sustained release tablets that release the active ingredients over 8-12 hours. Both product tablets are 0.500" round and 0.290" thick.
  AKG and AKG salts are grandfathered as GRAS compounds because these compounds were supplements prior to the Dietary Supplement Health and Education Act of 1994 ("DSHEA"). AKG and AKG salts are currently sold in the United States as supplements.
  The other components of the tablets are Vitamin A for the men's product and Vitamin D3 for the women's product. Vitamin A and Vitamin D are GRAS compounds per the FDA
  Arms: Females study product; Males study product
Dietary Supplement: Placebo — Matching placebo tablets are composed of Cellulose, Carnauba wax and/or rice bran wax (to match the specs), stearic acid, magnesium stearate and silica.
  Arms: Females placebo; Males placebo

SUMMARY:
In this randomized, double-blind, placebo-controlled trial in adult men ages 45-65 years and postmenopausal women to age 75 years, the anti-inflammatory property of proprietary CaAKG based dietary supplements will be assessed by the measurement of C-reactive protein (CRP) as the primary endpoint. Secondary safety endpoints will be assessed by monitoring blood chemistry results and recorded adverse effects. In addition, the biological age of the participants will be determined by the level of DNA methylation measured from saliva samples.

An open label Sub-Study was conducted on eligible and consenting subjects who were assigned to the placebo. Assessments and endpoints remained the same as for the main study.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled trial in adult men ages 45-65 years and postmenopausal women up to age 65 years to measure the effect that Rejuvant dietary supplement products have on inflammation by the measurement of C-Reactive Protein (CRP).

The study has four groups as outlined in Table 1. Groups 1-4 are divided by gender and each Group will receive the gender-specific investigational product or placebo.

Rejuvant and placebo tablets are 0.500" round and 0.290" thick. Groups 1 and 3 will take two tablets per day of the gender-specific investigational dietary supplement product. Groups 2 and 4 will take 2 placebo tablets per day. All Groups will take the investigational product for nine months. Participants will be assessed at four timepoints: Study Initiation (Day 1), Month 3, Month 6, and Month 9. At each visit weight, blood pressure, pulse, safety labs, CRP, blood chemistries, Hemoglobin A1C, and uric acid levels will be obtained, and the study questionnaire will be completed by each participant. These data will allow for an assessment of the antiinflammatory effects and the safety of the investigational dietary supplement products.

Additionally, up to 200 plasma metabolites will be measured. These data will be used to assess changes in participant metabolism over the course of the study. The blood chemistry and metabolite data may also be used to calculate the biological age of the participant by one or more published algorithms. DNA methylation analysis of saliva will determine the degree of DNA methylation (the cytosine of the CpG dinucleotide can be methylated). The degree of DNA methylation is correlated with aging and can be used as another measure of the biological age of the participant.

ELIGIBILITY:
Inclusion Criteria:

1. Men between the ages of 45 and 75 years
2. Postmenopausal Women up to age 75 years per EMR. Women should not have had a menstrual period for at least one year prior to enrollment into the study

Exclusion Criteria:

1. Diabetes as determined by the presence of EMR based diagnosis including prescribed any DM medications
2. Diagnosed with severe mental illness, substance abuse disorders per EMR
3. Diagnosed with congestive heart disease per EMR
4. Had a myocardial infarction in the previous year per EMR
5. EMR based Diagnosis of any Cancer in the past 5 years
6. EMR based diagnosis of morbid obesity or anorexia nervosa
7. Hospitalized in the previous 12 months
8. Active smoking

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Males 45 to 75 years old Postmenopausal Females up to age 75
Enrollment: 100 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Primary Outcome CRP, hs-CRP | 9 months
  The primary objective is to observe the effect, if any, of Rejuvant products on the C-reactive protein level (CRP, hs-CRP). These tests will be done at Day 1, Month 3, Month 6, and Month 9

SECONDARY OUTCOMES:
Safety Vital Signs | 9 months
  The secondary objective is to determine the safety of oral administration of Rejuvant products through assessments of height (Day 1 only), weight, blood pressure, heart rate, and temperature at Day 1, Month 3, Month 6, and Month 9 visits
Safety Laboratory Assessments | 9 months
  At Day 1, Month 3, Month 6, and Month 9 visits, laboratory assessments will be completed including Complete Blood Count, Comprehensive Metabolic Panel, and Lipid Panel
Additional Laboratory Tests | 9 months
  At Day 1, Month 3, Month 6, and Month 9 visits, laboratory assessments will be completed for Uric Acid and Hemoglobin A1C

OTHER OUTCOMES:
Metabolic Screen | 9 months
  Blood samples taken during site visits Day 1, Month 3, Month 6, and Month 9 will be tested and analyzed by an independent laboratory
Saliva Sample for DNA methylation analysis | 9 months
  Saliva samples will be obtained at the Day 1, Month 3, Month 6 and Month 9 visits. The saliva will be used for measurement of the degree of DNA methylation

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No